CLINICAL TRIAL: NCT05629897
Title: Randomised Clinical Trial to Evaluate the Efficacy of an Online Cognitive Rehabilitation Programme (COPERIA-COG) for Patients With Persistent COVID-19
Acronym: COPERIA-COG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Collaborators: Centro de Investigación Biomédica en Red de Salud Mental (Network); Galician South Health Research Institute (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COPERIA-COG
Record Dates: First submitted 2022-11-18; First posted 2022-11-29 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: COVID-19; Neuro-Degenerative Disease; Psychological; SARS CoV 2 Infection
Keywords: Cognitive rehabilitation; SARS-CoV-2; COVID; Long-term memory; Verbal learning; RAVLT
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Intervention or waiting list
Who Masked: Outcomes Assessor
Masking Description: The investigator performing the analysis will be blinded to which group is the active intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): They will perform an initial test of processing speed, attentional span and executive control. After this test, they will start the training programme. It consists of 40 sessions of cognitive stimulation, distributed over 8 weeks of treatment with a frequency of five sessions per week. In the last session, a final test will be performed, the same as the initial one.
  Interventions: Other: Sessions of cognitive stimulation
- Waiting list (No Intervention): They will perform an initial test of processing speed, attentional span and executive control. In the last session, 8 weeks after the initial test, a final test will be performed, the same as the initial one.
  They will have the opportunity to perform the same training as the experimental group after performing the final test. At 8 weeks, patients on the waiting list will be taught, if the wish, how to use the platform to perform the stimulation. They will be offered cognitive training with COPERIA-COG under the same conditions, periodicity, automatic reminders and calls from the psychologist as in the intervention group.

INTERVENTIONS:
Other: Sessions of cognitive stimulation — 40 sessions of cognitive stimulation of approximately 20 minutes duration per session are carried out, using the COPERIA platform.
  Arms: Intervention

SUMMARY:
The pandemic caused by SARS-CoV-2 infection has led to the emergence of diffuse and heterogeneous persistent symptoms in addition to the well-known acute symptoms, which have come to be referred to as persistent COVID. In particular, one of the frequent complaints of patients with a previous diagnosis of COVID is impaired cognitive ability.

Various cognitive rehabilitation programmes have benefited from incorporating the methodology of so-called "serious games" are designed to train or change behaviour while entertaining players. The design of the online rehabilitation programme (COPERIA-COG) took into account the principles of neuropsychological rehabilitation (neuropsychological pre-assessment, operational goal setting, task prioritisation and continuous feedback system) and combined different individual techniques, such as restitution and compensation. Patients treated with COPERIA-COG will show neuropsychological improvements in verbal memory compared to the waiting list group.

The main objective is to identify differences in long-term memory in patients treated with COPERIA-COG vs. patients on the waiting list. For this purpose, both groups will be evaluated through RAVLT, taking the long-term memory subtest as a reference, comparing the results before and after the active group performs the online training with COPERIA-COG.

The COPERIA platform is a cloud platform that provides a range of ICT tools for monitoring and aiding the recovery of patients with persistent COVID. To achieve this goal, the platform will store patient data to which Artificial Intelligence techniques will be applied to perform an assessment of the affected person.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤70 years old.
2. Read and write.
3. Diagnosis of persistent COVID according to WHO criteria.
4. The patient reports cognitive dysfunction with self-assessed impact of at least grade 2 on the Post-Covid Functional Status (Chile) (Klok et al., 2020, Lorca et al., 2021).
5. The patient does not present cognitive dysfunction to a degree equal to or greater than 1.5 SD assessed in the psychology consultation by means of the following instruments: RAVLT Rey Auditory Verbal Learning Test (Schmidt, 1996). Subtests of the Number Key, Symbol Search and Digit Span of the Scale for Measuring Adult and Adolescent Intelligence (WAIS III) (Wechsler, 1999). TMT Stroke Test (Reitan & Wolfson, 1993). Verbal fluency tests (Benton et al., 1989). In case of scores above 1.5 SD below the normative mean, they will be excluded from the study and referred for treatment to the Brain Injury Unit (Winblad et al., 2004).
6. Patients with capacity to consent and agree to participate in the study.
7. Patients who know how to use and have a Smartphone or Tablet and an Internet connection.

Exclusion Criteria:

1. Minors or persons legally incapacitated.
2. Previous neurological or psychiatric pathology involving neuropsychological compromise.
3. Active Covid19 infection.
4. Home oxygen therapy > 16 hours or home CPAP-BiPAP.
5. Be undergoing another cognitive rehabilitation process at the time of inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-12-14 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
RAVLT Rey Auditory Verbal Learning Test | 8 weeks
  An instrument that has proven useful in assessing verbal learning and memory. Easily administered test that assesses immediate memory span, new learning, susceptibility to interference and recognition memory.

SECONDARY OUTCOMES:
Subtests of the Number Key, Symbol Search and Digit Search Scale for Measuring Adult and Adolescent Intelligence (WAIS III) | 8 weeks
  They allow the calculation of the processing speed index. The Spanish adaptation of the WAIS-III was used. Reliability coefficients (two halves) range from .77 to .96.
Trail Making Test (TMT) | 8 weeks
  The test consists of two parts, A and B. Part A assesses sustained attention, processing speed, motor skills and visuospatial visual search skills. Part B assesses alternating attention and cognitive flexibility. Its reliability is between 0.86% and 0.94% and its reliability is .66. Neuronorm scales are used in Spain
Verbal fluency tests | 8 weeks
  The investigators will use the phonemic fluency test, a task of oral production of words before phonetic commands (P-M-R) and the semantic fluency test (animals), a task of linguistic production that requires the implementation of the mechanisms of access to the lexicon. Neuronorm scales are used in Spain. The scale is made with scalar scores from 2 to 18, where 2 is the worst score and 18 is the best.
Memory Failures Everyday-30 (MFE-30) | 8 weeks
  It is a 30-item questionnaire that explores the relationships between the occurrence of memory complaints, prefrontal symptomatology and perceived stress.
  The scale has values between 0-120. Where 120 is indicative of more severe impairment in daily functioning and 0 indicates optimal functioning.
Hospital Anxiety and Depression Scale (HADS Scale) | 8 weeks
  The Hospital Anxiety and Depression Scale was originally designed as a screening instrument for the detection of patients with affective disorders in response to the drawbacks of widely used instruments such as the GHQ. It consists of two sets of seven items -one representing the anxiety subscale and the other the depression subscale- both of which are psychopathological concepts of anxiety and depression independent.
  There are two subscales (anxiety and depression) with a score from 0 to 21 each. Scores greater than 10 are considered indicative of morbidity, scores between 8-10 are considered bordeline and scores less than 8 indicate no significant morbidity.
Adherence to online treatment | 8 weeks
  Number of games played and total time of use will be extracted from the platform, analysing whether there are differences by age or gender or severity.

OTHER OUTCOMES:
Age | 8 weeks
  Years
Sex | 8 weeks
  Male, Female
Level of education attained | 8 weeks
  School, High school, College, Superior
Employment status | 8 weeks
  Employed, unemployed, retired
Current treatment | 8 weeks
  Treatment taken by the patient at the time of the study.
Date of the SARS-CoV-2 PCR+ | 8 weeks
  DD-MMM-YYYY
Epidemic wave | 8 weeks
  Of the 7 waves of COVID-19 that have occurred in Spain, a description will be given of the wave to which the infection of each patient included belonged. First, second, third, fourth, fifth, sixth, seventh, eighth, ninth or tenth wave.
Vaccination status at the time of infection | 8 weeks
  Number of vaccine doses at the time of infection

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Galicia Sur Health Research Institute (IISGS) - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Complexo Hospitalario Universitario de Ourense, Ourense